# **Virginia Polytechnic Institute and State University**

# TOGETHER: A Couple's Model to Enhance Relationships and Economic Stability

**Unique Protocol ID: 15-960** 

**Consent Form** 

**Date: March 29, 2018** 

#### VIRGINIA POLYTECHNIC INSTITUTE AND STATE UNIVERSITY

**Informed Consent for Participants** in Research Projects Involving Human Subjects

Title of Project: TOGETHER: A Couples' Model to Enhance Relationships and Economic Stability

Investigator(s): Dr. Mariana Falconier <u>marianak@vt.edu</u> (703) 538 8461

Dr. Jinhee Kim <u>jinkim@umd.edu</u> (301) 405-3500

# I. Purpose of this Research Project

The main purposes of this project are to examine if the TOGETHER program is effective in improving couple relationships and economic stability and to evaluate the process of implementation of the program. The TOGETHER program includes a 20-hour comprehensive relationship and financial education workshop, case management for access to community resources and services, and opportunities for job and career advancement services if they are needed by participants. The project will enroll 720 study couples where partners are 18 and older, live together for at least 12 months, can communicate in English, live in Northern Virginia, Prince George's County, Maryland, or Montgomery County, Maryland, at least one partner is not retired, have no risk of domestic violence, feel safe participating with their partner in the program, do not have a current diagnosis of a severe psychiatric disorder that required hospitalization in the last 12 months, and have no cognitive impairment, or/and severe untreated substance abuse disorder. The program is open to both opposite and same-sex couples from any racial/ethnic or religious group.

In order to evaluate the program, a computer program will randomly assign half of the program couples (360 couples) in one group who will receive the TOGETHER Program and another half (360 couples) into another group who will not receive the program. Data from both groups will be compared to assess the effectiveness of the interventions. For such purposes, all couples will be completing surveys. The data from these surveys will be used to create reports for the funding agency, the Administration for Children and Families, and also to be published in academic articles and publications. However, your identifying information will never be included in any publications using the data.

This project is funded by the Department of Health and Human Services (HHS), Administration for Children and Families (ACF), Office of Family Assistance (OFA) under the Healthy Marriage and Responsible Fatherhood (HMRF) program (Grant Number: 90FM0077-01-00). The project is conducted in partnership with the University of Maryland, Family Services, Inc. (part of the Sheppard Pratt Health System), and the SkillSource Group, Inc.

#### II. Procedures

If both you and your partner agree to participate, both partners must consent and must first sign two copies of this form. One copy will be saved for the study team and one for you and your partner to keep. Consent from both partners is required for participation in the program. If one partner decides to withdraw, both partners will be withdrawn from the program because this program is designed for couples. After you sign the consent form, a case manager will meet with you and your partner

separately for 10 minutes. The case manager will ask questions that will help us determine whether it is safe for you and your partner to participate. If either partner reports feeling unsafe to participate with the other partner in this program and/or the case manager considers that it is not safe, you will not be allowed to participate and the case manager will refer you to appropriate domestic violence services. In cases of mild to moderate risk of domestic violence we may allow you to participate as long as you agree to participate in appropriate domestic violence services, you agree to authorize us to exchange information with the domestic violence agency about your situation, and/or you agree to sign a non-violence agreement with your partner. Following the screening interview for domestic violence, an automated computer system will decide whether you and your partner will be assigned to a group that will receive the TOGETHER program (INTERVENTION Group) or another group that will not (CONTROL Group). We cannot change the assignment of group. Once you are assigned to a group, we will ask your contact information for the intake. You will complete a short questionnaire about your demographic characteristics, financial well-being, and health on a tablet. The questionnaire is also available in paper format if you do not wish to complete it on the tablet. The questionnaire will take about 15 minutes. After this point, the procedure will be different whether you are assigned to the INTERVENTION or the CONTROL group. Two flowcharts showing the various steps for each group are provided for your information. Note that both, intervention and control groups, will complete the same Pre-Survey (initial), Post-Survey (8 weeks after the Pre-Test Survey), and Follow-up Survey (6 months after Post-Survey, which is the end of the program) and will receive the same incentives (gift cards) for their completion.

#### II. A. Participants Not Assigned to the TOGETHER Program (CONTROL Group)

Couples in this group will not participate in the TOGETHER program. Alternately, you and your partner will be invited to attend a three-hour Financial Literacy Workshop about 8 months after the enrollment in the program, at the time of completion of the Follow-up Survey. To evaluate our program, we will collect a series of surveys from you and your partner using tablets during our study. If the Internet is not working or if you prefer, you may complete the paper surveys. If you miss the meeting for the surveys, you will be mailed the surveys with instructions on how to complete them or be emailed with the instruction with the online survey link to complete them online when this option is available. You will complete the first survey called the Pre-Test Survey (90 minutes long) today. Your second survey called the Post-Test Survey (90 minutes long) will take place 8 weeks and your last survey called the Follow-Up Survey (90 minutes long) will be scheduled six months after the date of the Post-Test Survey. After you complete the Follow-up survey, you have the option of attending the three-hour Financial Literacy Workshop on the same day.

# II.B. Participants Assigned to the TOGETHER Program (INTERVENTION Group)

# **Outline of Program Activities**

Our programs are designed for couples therefore both you and your partner are expected to participate together in the program activities except for the job and career enhancement services for which only one of you may be in need of those services. You will be participating in the following program activities: (1) TOGETHER Workshop; (2) Case Management Meetings (in person or by phone); and (3) Job and Career Enhancement Services (as needed).

#### 1) **TOGETHER Workshop**:

- o 20-hour relationship and financial educational workshop
  - Nine modules that teach couples skills to improve:
    - Communication in general and about money problems in particular
    - Individual and couple coping in general and regarding financial stress
    - Problem-solving together as a couple
    - Financial management.
  - Consists of 8 sessions of 2 hours and 30 minutes each
    - Each session includes:
      - o A warm-up activity
      - o Brief review of past session content and homework
      - o Presentation and practice of new content
      - o Summary of all contents covered in the session
      - o Assignment of new homework
      - A 5-minute evaluation of the session and the homework
      - After each session, couples are assigned homework so that the skills learned in the session can be practiced between sessions.
  - Co-led by a couple expert and a financial expert
  - Each group has between 4 and 8 couples
- o Each session will take place at the same time and on the same day each week.
- You and your partner will be expected to attend the 8 sessions at either Family Services, Inc. or Virginia Tech, Falls Church, VA or other locations depending on your place of residence.
- o For the 1<sup>st</sup> session of the TOGETHER workshop you will be required to arrive 90 minutes earlier in order to complete a Pre-Test Survey on a tablet.
- o For the 8<sup>th</sup> session of the TOGETHER workshop, you will be asked to fill out a 90-minute Post-Test Survey on a tablet after the session ends.
- o If the Internet is not working or if you prefer, you may complete the paper surveys. If you miss the meeting for the surveys, you will be mailed the survey with detailed instructions or you may be given a link and individual passcode to complete them online if this option is available.
- Three months after you complete the TOGETHER workshop (all 8 sessions), you will be invited to attend a booster workshop session (3-hour) as a review of the TOGETHER workshop.
- The TOGETHER workshop that you were signed up for may be rescheduled if there are not enough participants.

#### 2) Case Management Meetings:

- You will be assigned a case manager at either Family Services, Inc.
  (Gaithersburg, MD), the University of Maryland, or the Women's Center
  (Vienna, VA) depending on your place of residence.
- You will have 7 meetings in total, as outlined below; held at the Women's Center, Virginia Tech, University of Maryland, Family Services, Inc., or by phone. A schedule of program participation will be provided for you.

#### • Intake and Enrolment Meeting (60 minutes):

- Assessment with you and your partner so that the areas where you or other household family members need assistance can be identified. The areas to be evaluated are housing, health, health coverage, transportation, mobility, food, substance abuse treatment, education, mental health treatment, legal issues, employment issues, child care, etc. If you are unable to stay for the Needs' Assessment, the case manager will schedule a meeting for another day with you and your partner or will offer the possibility to complete it by phone with both you at a later upon agreed day and time.
- O At the end of the meeting, you will be registered for the TOGETHER workshop and scheduled for the next 6 meetings with the case manager.

#### • Individual and Couple Development Plan Meeting (90 minutes):

- This meeting will take place 1-2 weeks after the Intake and Enrollment Meeting
- You and your partner will meet with your case manager to develop your individual and couples' long-term goals:
  - Agreeing on action steps
  - Establishing a timeline
  - Receiving referrals as part of your goals
- O Your case manager will discuss barriers and resources for the plan.
- The case manager will offer referrals as part of the action steps to meet your goals (i.e., housing, TANF, health care, child welfare, child support services, mental health services, and job and career enhancement services).
- If you are unable to attend this meeting in person, the case manager will schedule a phone meeting with you and your partners to complete the Individual and Couple Development Plan

#### • 5 Progress and 1 Exit Meeting (30 minutes each):

- o A meeting will occur every 5 weeks, during a period of 7 months
- o These meetings will start before you finish the TOGETHER workshop
- O Three of these meetings are suggested to be over the phone and three in person but they can all be over the phone if you and your partner cannot attend them in person.
- O You will meet with your case manager to:
  - Check progress towards goals established in the ICDP
  - Update the ICDP if necessary
  - Address barriers towards meeting ICDP goals
- Your final meeting with your case manager will be the exit meeting and will take place approximately 6 months following your last TOGETHER program workshop.
  - At the exit meeting, you will also fill out the Follow-up Survey for 90 minutes on a tablet after you complete the exit meeting. If the Internet is not working or if you prefer you can complete the paper survey. If you miss the meeting for the surveys, you will be mailed the survey with detailed instructions. You will evaluate the ICDP, future plans, and the program TOGETHER. This meeting will conclude your participation in the program.

#### 3) Employment Services (If Needed):

- For those who are looking for a job or wish to change or improve their work situation, you are invited to participate in job and career enhancement services.
- o This will be determined as a result of the Needs Assessment and will be incorporated into your Individual and Couple Development Plan.
- If you need such services, your case manager will make an appointment with an *employment case manager* at either the SkillSource Group, Inc., University of Maryland, or Family Services, Inc. to connect you to services in Virginia or Maryland depending on your place of residence.
- This appointment will be for a date immediately following the last session of the TOGETHER workshop.
- Your case manager will also ask you to sign an authorization to release information to the employment case manager about your Needs Assessment, Individual and Couple Development Plan, any concerning issues of safety, and any necessary information for the coordination of services.
  - However, the case manager should not disclose any confidential information about the couple beyond what is strictly necessary to coordinate services.
  - Releases may be rescinded by you and your partner any time.
- O At the employment agencies you will be given an overview of the services, eligibility criteria, responsibilities of participants, and agency policy. If you agree to receive services from the employment agency, you will be subjected to their terms and policies. The employment agency will see if you are eligible for any services they provide. If you are not eligible for the services they provide for free, we may pay for services for a period of six months starting from the day of the Post-Test Survey.
- Ouring the time that you participate in the present study we will request the employment agency to provide us with information on the Employment Individual Plan that they develop for you as well as the number and type of trainings and services that you receive. Once your participation in our study concludes, you may continue receiving services through the employment agency subject to their terms and policies.
- As part of the Intervention Group you may be invited to participate in a small group focus group discussion for 60 minutes (4 people per group). You will be asked about your experiences with the TOGETHER program, including your satisfaction with the program and our integration of services. This focus group will be conducted by the independent evaluator, AVAR consulting to maintain the objectivity of the evaluation.

#### III. Termination of Participation in the Study

Participation in the program concludes when you complete the Follow-up Survey, which takes place approximately 6 months after you completed the Post-Test Survey. However, you may be asked to discontinue program participation if such participation involves risks beyond the ones outlined in the present consent form. Such risks could include but are not limited to issues of domestic violence.

- If we consider that you and your partner are at risk of domestic violence from the initial screening or any subsequent meetings or interactions during the program, we may ask you not to continue in the program and may refer you and your partner to domestic violence services.
- In cases of mild to moderate risk of domestic violence, and as long as you and your partner consider that participation is safe for both of you, you may be allowed to continue to participate in the TOGETHER program. However, participation in domestic violence services may become a requirement for participation.

#### IV. Risks

#### IV.a. Participants Assigned to the TOGETHER program

The risks of participating in the TOGETHER program and completing program surveys are small. You might experience some uncomfortable feelings such as sadness or anger or conflict with your partner. You do not have to answer any questions or participate in any activities for the TOGETHER program that make you feel uncomfortable. If you would like to talk about your feelings or if you experience any conflict with your partner as results of participating in TOGETHER program activities or completing these surveys, please do the following.

- o (a) let program staff (case manager or workshop facilitators) know about you discomfort so that she/he can give you the name of a trained professional/ hospital/ crisis center, or, if you are in immediate danger
- o (b) call 911 or go to the nearest emergency room,
- o (c) call the county crisis hotline (Montgomery County 240-777-4000; Prince George's County 301-927-4500; Fairfax County 703-527-4077; Arlington County. 703-527-6603).

#### IV.b. Participants Not Assigned to the TOGETHER program

The risks of participating in the three-hour financial literacy workshop and completing surveys are very small. You might experience some uncomfortable feelings such as sadness or anger. You do not have to answer any questions that make you feel uncomfortable. You can stop at any time. If you would like to talk about your feelings or if you experience any conflict with your partner as a result of completing the workshop or surveys, please do the following.

- Let program staff (case manager or workshop facilitators) know about you discomfort so that she/he can give you the name of a trained professional/ hospital/ crisis center or, if you are in immediate danger.
- o Call 911 or go to the nearest emergency room.
- Call the county crisis hotline (Montgomery County 240-777-4000; Prince George's County 301-927-4500; Fairfax County 703-527-4077; Arlington County. 703-527-6603).

#### V. Benefits

#### V.a. Participants Assigned to the TOGETHER program

While we cannot promise that you will benefit from participating in this program, you might learn more about yourself and your relationship with your partner. Your participation in the TOGETHER Workshop, case management (access to community resources and services), and employment

services (opportunities for job and career advancement services) might help you improve your couple relationship, stress management skills, financial management skills, and economic stability. This improvement might help you deal with economic difficulties in a way that is not destructive to you and/or to your couple's relationship. In addition, the information you share through the surveys and your participation in the TOGETHER program may help improve TOGETHER and other healthy marriage programs that may benefit other couples through improved understanding of couple relationships and economic stability.

## V.b. Participants Not Assigned to the TOGETHER program

While we cannot promise that you will benefit from participating in the financial literacy workshop and completing surveys, you might learn more about financial management and, to some extent, to your couple's relationship as well. In addition, the information you share with the program staff through the surveys will help improve the TOGETHER program and other healthy marriage programs that may benefit couples in the future.

# VI. Extent of Anonymity and Confidentiality

Your participation in this program will be kept confidential by the program staff including case managers and facilitators.

- During the TOGETHER workshop, you can use a pseudonym. You will not be forced to reveal your real identity if you do not wish to do so.
- All information you share verbally, in writing, or electronically through surveys during your participation in the TOGETHER program will not be disclosed to any individuals outside the research team. No one, except the program staff members, will see or hear your answers.
- All information collected during this program and recorded in paper format will be stored in a locked file cabinet in a locked office. Only members of the program staff will be able to open the office and file cabinet.
- An electronic database containing only your answers to the surveys will be kept for future use, but only designated program staff (including our independent evaluator AVAR Consulting) will have access to this database. This database will not contain any personally identifiable information, and it will be securely protected.
- Results of this study may be used in reports, publications and presentations. However, we will not include any identifiable information. Your study data will be handled as confidentially as possible. If results of this study are published or presented, identifiable information will not be used.
- The funding Agency, the Office of Family Assistance in the Administration of Children and Families, U.S. Department of Health and Human Services (HHS), Administration for Children and Families have access to your data including identifying information via their online data management system called nFORM. The system is consistent with the Privacy Act, the Health Insurance Portability and Accountability Act, the Federal Information Security Management Act, and National Institute of Standards and Technology security and privacy standards.
- Identifiable data will be encrypted at all times (in transit and at rest) using cryptographic modules that are compliant with Federal Information Processing Standard 140-2, and will be securely deleted from the system when no longer needed.

- The first part of the surveys that you will be completing (Applicant Characteristics/ Demographic Information, Pre-Test, and Post-Test) will be entered into the nFORM system.
  - You will be informed for each of these surveys where the section that is entered in the nFORM system starts and ends.
  - The Follow-up Survey is not entered in nFORM. None of the surveys in the nFORM system contain personal identifying information but an identification number.
  - However, nFORM will keep a file for you and your partner with personal identifying information and the services that you are receiving through the TOGETHER program.
- The Virginia Tech (VT) Institutional Review Board (IRB) may view the study's data for auditing purposes. The IRB is responsible for the oversight of the protection of human subjects involved in research.
- We will protect your confidentiality unless we think you are a threat to yourself or someone else and in cases of suspected child abuse or neglect, in which cases we must report the situation to the appropriate government authorities. That is the only time in which your confidentiality would not be protected.

## VII. Compensation

We cannot fully repay you for your time and effort but we provide gift cards as a token of our appreciation. Compensation will be different depending upon your group assignment.

- CONTROL and INTERVENTION groups will receive gift cards for the completion of the Pre-Test, Post-Test, and Follow-Up Surveys when both partners have completed the surveys. You will be reimbursed as follows:
  - a. A \$20 gift card for each partner after completion of Pre-Test Survey
  - b. A \$20 gift card for each partner after completion of Post-Test Survey
  - c. A \$40 gift card for each partner after completion of survey at 6 months follow-up
- In the INTERVENTION couples group each partner will receive a \$20 gift card for their participation in the Individual and Couple Development plan meeting with the case manager and the following gift cards depending on their level of attendance to the TOGETHER workshop (presented in the3<sup>rd</sup> Progress meeting by the case manager after attendance is verified)
  - a. A \$40 gift card for each partner if both partners have attended the 8 sessions
  - b. A \$30 gift card for each partner if both partners have attended the 7 sessions
  - c. A \$15 gift card for each partner if both partners have attended the 6 sessions.
- In the INTERVENTION couples group we will provide childcare support (up to \$280) if you have children ages below 12 and need child care to participate in the program whenever child care support is not provided for free at the site or a nearby location where the TOGETHER workshop session are offered. In order for your licensed care provider to be reimbursed, we will ask you to have your provider complete a W-9 for tax reporting, the Child Reimbursement forms, and obtain the signature of the licensed childcare provider.

Virginia Tech requires that any gift amount received over \$75 is considered taxable for each of you and therefore, Virginia participants will be asked to fill out the corresponding IRS forms regardless of whether you reside in Virginia or in Maryland. Maryland participants will be asked to fill out the Social Security Form only when they are Intervention Group (total gift amount will exceed \$100 per person).

The funding agency for the present study, Administration for Children and Families (ACF), U.S. Department of Health and Human Services requires the following restrictions on the use of gift: cards cannot be redeemed for cash, transferred to third parties, or used to purchase entertainment, alcohol, tobacco, or firearms. Your voluntary participation in this study is also an indication that you will conform with the restrictions established by the sponsor. If you do not want to accept those restrictions, then you should not participate in the study.

#### VIII. Freedom to Withdraw

Participation in this study is entirely voluntary. You have the right to leave the study at any time without penalty. You can withdraw your consent to participate in this program at any time. We also can provide a form for you to withdraw from the program. However, since the TOGETHER program has been designed to assist couples and many of the activities involve both members of the couple, if you decide to withdraw, both you and your partner will withdraw from the study. Should you withdraw or otherwise discontinue participation, you will be compensated for the portion of the project completed in accordance with the Compensation section of this document. While you are participating in the TOGETHER program activities or answering surveys or questions, you are free not to answer any questions that you choose or respond to what is being asked of you without penalty.

#### IX. Questions or Concerns

Should you have any questions about this study, you may contact one of the research investigators whose contact information is included at the beginning of this document.

Should you have any questions or concerns about the study's conduct or your rights as a research participant, or need to report a research-related injury or event, you may contact the Virginia Tech Institutional Review Board at irb@vt.edu or (540) 231-3732.

In addition, if you are a Maryland resident, are receiving services through Family Services, Inc. (part of Sheppard Pratt Health System, ad have questions regarding your rights as a research participant you may contact Dr Faith Dickerson of the Sheppard Pratt IRB at 410-938-3000.

#### X. Subject's Consent

| I have read the Consent Form and conditions of this project. I have had all my questions answered |
|---|
| hereby acknowledge the above and give my voluntary consent: |

| | Date |
|-----------|------|
| Signature | |

Printed name